CLINICAL TRIAL: NCT02936596
Title: Biochemical Response of Primary Biliary Cholangitis-autoimmune Hepatitis Overlap Syndrome Induced by Ursodeoxycholic Acid Only or Combination Therapy of Immunosuppressive Agents
Brief Title: Remission Induction of Primary Biliary Cholangitis-autoimmune Hepatitis Overlap Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiaoli Fan (Other)
Responsible Party: Sponsor-Investigator, Xiaoli Fan, Master Degree, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OS-1
Record Dates: First submitted 2016-10-15; First posted 2016-10-18 (Estimated); Last update posted 2021-10-27 (Actual); Status verified 2021-05

CONDITIONS: Hepatitis, Autoimmune; Cholangitis; Liver Cirrhosis, Biliary; Cholestasis
MeSH Terms: conditions — Hepatitis, Autoimmune; Cholangitis; Liver Cirrhosis, Biliary; Cholestasis | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ursodeoxycholic acid + immunosuppressive agents group (Experimental): Ursodeoxycholic acid + immunosuppressive agents
  Interventions: Drug: Ursodeoxycholic acid combination of immunosuppressive agents
- Ursodeoxycholic acid group (Active Comparator): Ursodeoxycholic acid
  Interventions: Drug: Ursodeoxycholic Acid

INTERVENTIONS:
Drug: Ursodeoxycholic acid combination of immunosuppressive agents — Ursodeoxycholic acid combination of immunosuppressive agents(methylprednisolone with or without azathioprine)
  Arms: Ursodeoxycholic acid + immunosuppressive agents group
Drug: Ursodeoxycholic Acid — Ursodeoxycholic Acid
  Arms: Ursodeoxycholic acid group

SUMMARY:
Biochemical response of primary biliary cholangitis-autoimmune hepatitis overlap syndrome induced by ursodeoxycholic acid only or combination therapy of immunosuppressive agents

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients aged 18-70 years;
* 2.Diagnosed with primary biliary cholangitis-autoimmune hepatitis overlap syndrome according to Paris criteria, based on liver biopsy results obtained 3 months before screening;
* 3.White blood cell count ≥2.5x10^9/L or platelet count ≥50x10^9/L at inclusion;
* 4.Agreed to participate in the trial, and assigned informed consent.

Exclusion Criteria:

* 1. The presence of hepatitis A, B, C, D, or E virus infection;
* 2. Patients with indications for immunosuppressive treatment at inclusion: serum alanine transaminase(ALT) or aspartate transaminase(AST) ≥10 fold upper limit of normal(ULN)，or serum ALT or AST≥ 5 fold ULN and γglobulin level ≥ 2 fold ULN, or bridging necrosis or multiacinar necrosis on histological examination.
* 3. Patients with complications of cirrhosis;
* 4. Patients with previous treatment of immunosuppressive agents or traditional Chinese medicine for more than one month;
* 5. Primary sclerosing cholangitis,non-alcoholic steatohepatitis,drug induced liver disease or Wilson's disease confirmed by liver biopsy;
* 6. Pregnant and breeding women;
* 7. Severe disorders of other vital organs, such as severe heart failure, cancer;
* 8. Parenteral administration of blood or blood products within 6 months before screening;
* 9. Recent treatment with drugs having known liver toxicity;
* 10.Taken part in other clinic trials within 6 months before screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2016-12; Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Percent of patients that achieve biochemical remission of autoimmune hepatitis(AIH) | Month 6 during treatment with ursodeoxycholic acid only or combination therapy of immunosuppressive agents

SECONDARY OUTCOMES:
Alanine transaminase (ALT) | Week 2 and Month 1, 3, 6
Aspartate transaminase(AST) | Week 2 and Month 1, 3, 6
Immunoglobulin G(IgG) | Week 2 and Month 1, 3, 6
Globin(GLB) | Week 2 and Month 1, 3, 6
Total bilirubin(TB) | Week 2 and Month 1, 3, 6
Direct bilirubin(DB) | Week 2 and Month 1, 3, 6
Alkaline phosphatase(ALP) | Week 2 and Month 1, 3, 6
Glutamyltransferase(GGT) | Week 2 and Month 1, 3, 6
Side effects | Evaluation of side effects during the study period(6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Li Yang, MD, Study Chair — West China Hospital,Chengdu, Sichuan, China
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided